CLINICAL TRIAL: NCT02110056
Title: Modulation of Visual-Spatial Learning in Healthy Older Adults by Transcranial Direct Current Stimulation - Proof of Principle and Mechanisms
Brief Title: Modulation of Visual-Spatial Learning in Healthy Older Adults by tDCS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Agnes Flöel, Prof. Dr., Charite University, Berlin, Germany
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: LOCATO-OA-tDCS
Record Dates: First submitted 2014-02-13; First posted 2014-04-10 (Estimated); Last update posted 2018-01-30 (Actual); Status verified 2018-01

CONDITIONS: Healthy Older Adults
Keywords: healthy older adults; tDCS; LOCATO task; visual-spatial learning
MeSH Terms: interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- training + tDCS (Experimental): Combination of intensive training of visual-spatial abilities (LOCATO task) with transcranial direct current stimulation (tDCS)
  Interventions: Device: tDCS; Behavioral: training
- training + sham stimulation (Sham Comparator): Combination of intensive training of visual-spatial abilities (LOCATO task) with sham stimulation
  Interventions: Device: tDCS; Behavioral: training

INTERVENTIONS:
Device: tDCS — transcranial direct current stimulation (tDCS)
Behavioral: training — intensive training of visual-spatial abilities (in LOCATO task)

SUMMARY:
The aim of this study is to investigate whether a combination of intensive training of visual-spatial abilities (LOCATO task) with anodal transcranial direct current stimulation (tDCS) leads to an improvement of learning and memory in healthy older adults and to examine the underlying neuronal mechanism.

ELIGIBILITY:
Inclusion Criteria (old healthy controls):

* right handedness
* unobtrusive neuropsychological screening
* age: 50-90 years

Exclusion Criteria:

* severe internal or psychiatric disease
* epilepsy
* other severe neurological diseases, e.g. previous major stroke or brain tumor
* DMS-IV manifest dementia
* contraindication for MRT (claustrophobia, metallic implants, tattoos)

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2014-03; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Performance in LOCATO task (Visual-Spatial learning and memory) after a combination of intensive visual-spatial training and tDCS | immediately after the end of a 3 day training period in tDCS condition compared to sham condition
  Investigation whether the combination of intensive visual-spatial training (LOCATO task) and tDCS leads to an improvement of visual-spatial learning and memory measured by performance in LOCATO task after end of a 3 day training period compared to sham stimulation.

SECONDARY OUTCOMES:
long term effects | after 1 month vs baseline
  long term effects measured by performance in LOCATO task after end of training and after 1 month compared to control condition
functional changes: Connectivity | after end of 3-day period of training vs baseline
  Connectivity (measured by resting-state fMRT and correlation analysis) at baseline compared to end of 3 day period of training
cortical excitability | at baseline
  measured by transcranial magnetic stimulation (TMS) at baseline
Quality of life | after 1 month vs baseline
  quality of life as measured by standardized questionaire at baseline compared to quality of life measured 1 month after intervention (training and stimulation vs. training and sham-stimualtion)
memory | immediately after end of 3-day of cognitive training, after 1 month vs. baseline
  memory performance tested at baseline compared to memory performance after the end of a 3-day cognitive training period and after 1 month (posttraining) in training and stimulation vs. training and sham stimulation
affective state | immediately after the end of 3-day cognitive training, after 1 month vs. baseline
  affective state measured at baseline compared to affective state measured after the end of a 3-day cognitve training period and after 1 month (posttraining) in training and stimulation vs. training and sham stimulation
genotyping of learning related polymorphisms | once
  To assess predictors of positive reaction to brain stimulation, genotyping of several learning related polymorphisms will be performed (i.e., APOE, BDNF Val66Met, COMT Val158Met).

CONTACTS AND LOCATIONS:
Overall Officials: Agnes Flöel, Prof. Dr., Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- Charite Universitätsmedizin Berlin, Berlin, Germany

REFERENCES:
- [Result] Antonenko D, Kulzow N, Cesarz ME, Schindler K, Grittner U, Floel A. Hippocampal Pathway Plasticity Is Associated with the Ability to Form Novel Memories in Older Adults. Front Aging Neurosci. 2016 Mar 22;8:61. doi: 10.3389/fnagi.2016.00061. eCollection 2016. PMID 27047376
- [Result] Antonenko D, Kulzow N, Sousa A, Prehn K, Grittner U, Floel A. Neuronal and behavioral effects of multi-day brain stimulation and memory training. Neurobiol Aging. 2018 Jan;61:245-254. doi: 10.1016/j.neurobiolaging.2017.09.017. Epub 2017 Sep 28. PMID 29050849